CLINICAL TRIAL: NCT02346838
Title: The Effect of Prebiotics on Insulin Sensitivity, Metabolic Flexibility, and Cardiovascular Health in Prediabetic Adults.
Brief Title: Prebiotics, Gut Microbiota, and Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Kevin Davy, Kevin P. Davy, PhD, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Prebiotics-Prediabetes
Record Dates: First submitted 2015-01-07; First posted 2015-01-27 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Prediabetes
Keywords: Prediabetes, prebiotics, metabolic endotoxemia
MeSH Terms: conditions — Prediabetic State | interventions — Inulin; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inulin (Experimental): Participants will receive 10 g of inulin powder each day for 6 weeks.
  Interventions: Dietary Supplement: Inulin
- Placebo (Placebo Comparator): Participants will receive 10 g of maltodextrin each day for 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin — The treatment will be mixed in orange juice or other beverage and will be consumed at breakfast each day in our metabolic kitchen.
  Other Names: Prebiotic
  Arms: Inulin
Dietary Supplement: Placebo — The placebo will be mixed in orange juice or other beverage and will be consumed at breakfast each day in our metabolic kitchen.
  Arms: Placebo

SUMMARY:
Forty-eight prediabetic men and women (50-75 years of age) will participate in a 6-week feeding study in which they will randomized to receive either 10 g/day of inulin or placebo. All subjects will be fed an isocaloric diet (50% carbohydrate, 35% fat, 15% protein,) controlled for micronutrient content for 6 weeks to avoid the potential confound of individual differences in diet on gut microbiota. Measurements of intestinal permeability, insulin sensitivity, and skeletal muscle metabolic flexibility will be made prior to and following the controlled feeding period. Stool samples will be collected to assess gut microbial communities.

DETAILED DESCRIPTION:
Prebiotics have been defined as "selectively fermented ingredients that result in specific changes in the composition and/or activity of the gastrointestinal microbiota, thus conferring health benefit(s) upon host health". Commonly used prebiotics are inulin-type fructans, fructo-oligosaccharides, xylo-oligosaccharides and galacto-oligosaccharides and while all prebiotics are fibers, not all fibers are prebiotics. The proliferation of a targeted bacterial species, in particular, Bifiodobacterium spp. and Lactobacillus spp. contribute to host cardiometabolic health in many ways including, but not limited to, short chain fatty acid production and, modulation of gut barrier function, endotoxin concentrations, inflammatory pathways, and energy metabolism however, to our knowledge the potential benefits of prebiotic supplementation on cardiometabolic dysfunction has received little attention. Although the concept that dysbiosis of the gut microbiota leads to metabolic endotoxemia and increased risk of cardiometabolic disease is novel, very little information is available in humans. The significance of our proposal includes providing proof of concept efficacy of prebiotic supplementation with inulin on cardiometabolic dysfunction and assessing its relation with changes in gut bacterial communities, intestinal permeability, and metabolic endotoxemia in prediabetes, a condition affecting a substantial segment of the population. Our study could lead to the identification of prebiotic supplementation with inulin as a simple and efficacious strategy for reducing cardiometabolic risk in prediabetes which could change clinical practice by informing dietary recommendations and increasing acceptance of prebiotics by the scientific and medical community.

ELIGIBILITY:
Inclusion Criteria:

* Men and women; postmenopausal women not taking hormone replacement therapy.
* Fasting glucose between 5.6 - 6.9 mmol/L and/or a 2h plasma glucose between 7.8-11.1 mmol/L following a 75 g oral glucose tolerance test.
* Weight stable for previous 6 months (+/- 2.0 kg).
* Sedentary to recreationally active
* Willing to be randomized to treatment or placebo.
* Verbal and written informed consent.
* No plans to gain/lose weight or change physical activity level.
* Willing to pick up food daily, and consume foods provided for the 6-week controlled feeding period.

Exclusion Criteria:

* BMI less than 25 kg/m2 or greater than 40 kg/m2 or body mass greater than 300 pounds due to limit of DEXA.
* Diabetes or diabetes medications
* Prebiotic or probiotic supplement or product consumption in prior 3 months.
* Total cholesterol > 6.2 mmol/L; triglycerides > 4.5 mmol/L.
* Blood pressure > 140/90 mmHg or antihypertensive medications.
* Diagnosed inflammatory disease (e.g. lupus, irritable bowel, periodontal disease, etc)
* Fructo, galacto-, xylo-oligosaccharide intake > 3 g/day.
* Past or current ischemic heart disease, stroke, respiratory disease, endocrine or metabolic disease, neurological disease, or hematological-oncological disease.
* Smoking, alcohol consumption > 2 servings /d for males and 1 serving/d for females, or taking medications (including but not limited to statins or other drugs with anti-inflammatory actions) or antioxidant vitamins or supplements.
* Known allergy, hypersensitivity, or intolerance to inulin.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity. | Baseline, 6 weeks
  Insulin sensitivity will be assessed via a frequently sampled intravenous glucose tolerance test.

SECONDARY OUTCOMES:
Change in metabolic flexibility. | Baseline, 6 weeks
  Metabolic flexibility will be measured in skeletal muscle biopsies prior to and 4 hours following a high fat meal.
Change in endothelial function. | Baseline, 6 weeks
  Flow mediated dilation of the brachial artery will be assessed using duplex ultrasonography with a high resolution linear array transducer according to published guidelines.
Change in arterial stiffness. | Baseline, 6 weeks
  Arterial stiffness will be measured via carotid femoral pulse wave velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Davy, PhD, Principal Investigator — Virginia Polytechnic and State University
Locations (1):
- Virginia Polytechnic and State University, Blacksburg, Virginia, United States